CLINICAL TRIAL: NCT00522652
Title: A Phase 1 Trial of Oral PX-478 (a HIF-1α Inhibitor) in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Phase I Trial of PX-478
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Larry Romel / Sr. Director, Clinical Operations, Oncothyreon Inc
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-478-001
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2010-05

CONDITIONS: Advanced Solid Tumors; Lymphoma
Keywords: cancer; advanced cancer; lymphoma
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — 2-amino-3-(4'-N,N-bis(2-chloroethyl)amino)phenylpropionic acid N-oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Drug (Experimental): Dose Escalation
  Interventions: Drug: PX-478

INTERVENTIONS:
Drug: PX-478 — Oral formulation, dose escalation, taken on days 1 to 5 of a 21 day cycle until progression or development of unacceptable toxicity

SUMMARY:
This study is being conducted to determine the safety and biologic activity of PX-478, and to allow for observation of any preliminary evidence of antitumor activity in patients with advanced metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed the informed consent and must be considered legally capable of providing his or her own consent for participation in this study.
* The patient has a histologically or cytologically confirmed diagnosis of advanced solid tumor or lymphoma and has failed or is intolerant of standard therapy.
* The patient is ≥18 years of age.
* ECOG performance status 0 to 1.
* The patient has a predicted life expectancy of at least 12 weeks.
* Patients must have discontinued prior chemotherapy or other investigational agents for at least three weeks prior to receiving the first dose of study drug (six weeks for mitomycin C, nitrosureas, vaccines, or antibody therapy) and recovered from the toxic effects of that treatment (recovered to baseline or ≤Common Toxicity Criteria for Adverse Events (CTCAE) grade 1).
* Patients must have discontinued any radiation therapy at least four weeks prior to entry into the study and have recovered from all radiation-related toxicities (recovered to baseline or ≤CTCAE grade 1).
* The patient has adequate hematologic function defined as: WBC count >3,000 cells/μL; platelets >100,000/μL; hemoglobin >9 g/dL (may be transfused to this level); ANC >1500 cells/μL.
* The patient has adequate hepatic function defined as: bilirubin <1.5 mg/dL; aspartate aminotransaminase (AST/SGOT) & alanine aminotransferase (ALT/SGPT) <2.5 x ULN or <5 x ULN if due to metastatic disease.
* The patient has adequate renal function as defined by serum creatinine level <1.5 mg/dL.
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method; abstinence) prior to study entry and for the duration of study participation. The patient, if a man, agrees to use effective contraception or abstinence.

Exclusion Criteria:

* Patients with any active infection requiring i.v. antibiotics at study entry.
* Any serious concomitant systemic disorders that in the opinion of the investigator would place the patient at excessive or unacceptable risk of toxicity.
* Surgery within the four weeks prior to the first dose of PX 478.
* Significant central nervous system (CNS) or psychiatric disorder(s) that preclude the ability of the patient to provide informed consent.
* Known or suspected brain metastases that have not received adequate therapy. In the case of previously treated brain metastases, a minimum of four weeks interval between completion of radiation therapy and registration on study with radiologic evidence of stable or responding brain metastases is required. In the setting of previous CNS metastasectomy, adequate (minimum four week) recovery from surgery and/or radiation therapy should be documented.
* Patients with a history of seizures, non-healing wounds, or arterial thrombosis.
* Patients with unstable atrial or ventricular arrhythmias requiring control by medication; any cardiac ischemic event experienced within the preceding six months; prior history of congestive heart failure requiring therapy.
* Patients who are breastfeeding or pregnant (confirmed by serum β-HCG within 10 days prior to the start of study treatment if applicable).
* Patients with total gastrectomy or partial bowel obstruction.
* Any condition that could jeopardize the safety of the patient and compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the MTD of PX-478 administered orally on days one to five of a 21 day cycle | 21 days

SECONDARY OUTCOMES:
To evaluate the safety profile of PX-478 when administered orally on days one to five of a 21 day cycle | 42 days
To evaluate pharmacodynamic measures of the effects of PX 478 on the HIF 1-alpha pathway, and related tumor markers | 42 days
To determine the PK profile of PX 478 when administered orally on days one to five of a 21 day cycle | 21 days
To evaluate the effects of PX 478 on tumor blood flow and vascular permeability as measured by DCE MRI | 21 days
To evaluate the anti-tumor activity of PX 478 in patients with advanced malignancies | 42 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Palayoor ST, Mitchell JB, Cerna D, Degraff W, John-Aryankalayil M, Coleman CN. PX-478, an inhibitor of hypoxia-inducible factor-1alpha, enhances radiosensitivity of prostate carcinoma cells. Int J Cancer. 2008 Nov 15;123(10):2430-7. doi: 10.1002/ijc.23807. PMID 18729192